CLINICAL TRIAL: NCT04331795
Title: Early Institution of Tocilizumab Titration in Non-Critical Hospitalized COVID-19 Pneumonitis
Brief Title: Tocilizumab to Prevent Clinical Decompensation in Hospitalized, Non-critically Ill Patients With COVID-19 Pneumonitis
Acronym: COVIDOSE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB20-0515
Record Dates: First submitted 2020-04-01; First posted 2020-04-02 (Actual); Results first posted 2022-06-09 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — tocilizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Hospitalized, non-critically ill patients with COVID-19 pneumonitis with risk factors for decompensation
  Interventions: Drug: Tocilizumab
- Group B (Experimental): Hospitalized, non-critically ill patients with COVID-19 pneumonitis without risk factors for decompensation
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — Group A: Tocilizumab (beginning dose 200mg) Single dose is provisioned, patient is eligible to receive up to two doses, with re-evaluation of clinical and biochemical responses performed every 24 hours.
  Second dose is provisioned if:
  1. Increasing supplemental oxygen requirement or Tmax higher than baseline in the 24h following initial tocilizumab administration AND
  2. CRP decrease is < 25% at 24 hours following tocilizumab administration and CRP > 40mg/L
  Arms: Group A
Drug: Tocilizumab — Group B: Low-dose tocilizumab (beginning dose 80mg) Single dose is provisioned, patient is eligible to receive up to two doses, with re-evaluation of clinical and biochemical responses performed every 24 hours.
  Second dose is provisioned if:
  1. Increasing supplemental oxygen requirement or Tmax higher than baseline in the 24h following initial tocilizumab administration AND
  2. CRP decrease is < 25% at 24 hours following tocilizumab administration and CRP > 40mg/L
  Arms: Group B

SUMMARY:
Coronavirus disease-2019 (COVID-19) has a quoted inpatient mortality as high as 25%. This high mortality may be driven by hyperinflammation resembling cytokine release syndrome (CRS), offering the hope that therapies targeting the interleukin-6 (IL-6) axis therapies commonly used to treat CRS can be used to reduce COVID-19 mortality. Retrospective analysis of severe to critical COVID-19 patients receiving tocilizumab demonstrated that the majority of patients had rapid resolution (i.e., within 24-72 hours following administration) of both clinical and biochemical signs (fever and CRP, respectively) of hyperinflammation with only a single tocilizumab dose.

Hypotheses:

1. Tocilizumab is effective in decreasing signs, symptoms, and laboratory evidence of COVID-19 pneumonitis in hospitalized, non-critically ill patients with clinical risk factors for clinical decompensation, intensive care utilization, and death.
2. Low-dose tocilizumab is effective in decreasing signs, symptoms, and laboratory evidence of COVID-19 pneumonitis in hospitalized, non-critically ill patients with and without clinical risk factors for clinical decompensation, intensive care utilization, and death.

Objectives:

1. To establish proof of concept that tocilizumab is effective in decreasing signs, symptoms, and laboratory evidence of COVID-19 pneumonitis in hospitalized, non-critically ill patients with clinical risk factors for clinical decompensation, intensive care utilization, and death, as determined by the clinical outcome of resolution of fever and the biochemical outcome measures of time to CRP normalization for the individual patient and the rate of patients whose CRP normalize.
2. To establish proof of concept that low-dose tocilizumab is effective in decreasing signs, symptoms, and laboratory evidence of COVID-19 pneumonitis in hospitalized, non-critically ill patients without clinical risk factors for clinical decompensation, intensive care utilization, and death, as determined by the clinical outcome of resolution of fever and the biochemical outcome measures of time to CRP normalization for the individual patient and the rate of patients whose CRP normalize.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years of age
* Approval from the patient's primary service
* Admitted as an inpatient to University of Chicago Medicine
* Fever, documented in electronic medical record and defined as: T ≥ 38*C by any conventional clinical method (forehead, tympanic, oral, axillary, rectal)
* Positive test for active SARS-CoV-2 infection
* Radiographic evidence of infiltrates on chest radiograph (CXR) or computed tomography (CT)
* Ability to provide written informed consent on the part of the subject or, in the absence of decisional capacity of the subject, an appropriate surrogate (e.g. a legally authorized representative).

Exclusion Criteria:

* Concurrent use of invasive mechanical ventilation (patients receiving non-invasive mechanical ventilation [CPAP, BiPap, HHFNC] are eligible)
* Concurrent use of vasopressor or inotropic medications
* Previous receipt of tocilizumab or another anti-IL6R or IL-6 inhibitor.
* Known history of hypersensitivity to tocilizumab.
* Patients who are actively being considered for a study of an antiviral agent that would potentially exclude concurrent enrollment on this study.
* Patients actively receiving an investigational antiviral agent in the context of a clinical research study.
* Diagnosis of end-stage liver disease or listed for liver transplant.
* Elevation of AST or ALT in excess of 5 times the upper limit of normal.
* Neutropenia (Absolute neutrophil count < 500/uL).
* Thrombocytopenia (Platelets < 50,000/uL).
* On active therapy with a biologic immunosuppressive agent, which include the following biologics and any biosimilar versions thereof:
* Alemtuzumab
* Blinatumomab
* Brentuximab
* Daratumumab
* Elotuzumab
* Ibritumomab
* Obinutuzumab
* Ofatumumab
* Ocrelizumab
* Rituximab
* Inotuzumab
* Gemtuzumab
* Tositumumab
* Moxetumomab
* Polatuzumab
* Abatacept
* Adalimumab
* Belimumab
* Certolizumab
* Eculizumab
* Etanercept
* Golimumab
* Infliximab
* Ixekizumab
* Rituximab
* Sarilumab
* Secukinumab
* Tocilizumab
* Ustekinumab
* On active therapy with a JAK2-targeted agent, which include the following:
* Tofacitinib
* Baricitinib
* Upadacitinib
* Ruxolitinib
* History of bone marrow transplantation or solid organ transplant.
* Known history of Hepatitis B or Hepatitis C.
* Known history of mycobacterium tuberculosis infection at risk for reactivation.
* Known history of gastrointestinal perforation or active diverticulitis.
* Multi-organ failure as determined by primary treating team
* Any other documented serious, active infection besides COVID-19.
* Pregnant patients
* Patients who are unable to discontinue scheduled antipyretic medications, either as monotherapy (e.g., acetaminophen or ibuprofen [aspirin is acceptable]) or as part of combination therapy (e.g., hydrocodone/acetaminophen, aspirin/acetaminophen/caffeine [Excedrin®])
* CRP < 40 mg/L (or ug/mL)

Patients will be assigned to Group A if:

● C-reactive protein (CRP) ≥ 75 ug/mL

AND

Any one of the following criteria are met:

* Previous ICU admission
* Previous non-elective intubation
* Admission for heart failure exacerbation within the past 12 months
* History of percutaneous coronary intervention (PCI)
* History of coronary artery bypass graft (CABG) surgery
* Diagnosis of pulmonary hypertension
* Baseline requirement for supplemental O2
* Diagnosis of interstitial lung disease (ILD)
* Admission for chronic obstructive pulmonary disease (COPD) exacerbation within the past 12 months
* Asthma with use of daily inhaled corticosteroid
* History of pneumonectomy or lobectomy
* History of radiation therapy to the lung
* History of HIV
* Cancer of any stage and receiving active treatment (excluding hormonal therapy)
* Any history of diagnosed immunodeficiency
* End-stage renal disease (ESRD) requiring peritoneal or hemodialysis
* History of cerebrovascular accident with residual, patient-reported neurologic deficit
* BMI >30 kg/m2
* Supplemental O2 requirement > 6L in the 24 hours prior to enrollment and tocilizumab administration

All other eligible patients assigned to Group B

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-04-04 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2020-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pankti Reid, MD, MPH, Principal Investigator — University of Chicago, Department of Medicine, Section of Rheumatology
Locations (1):
- University of Chicago Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Strohbehn GW, Heiss BL, Rouhani SJ, Trujillo JA, Yu J, Kacew AJ, Higgs EF, Bloodworth JC, Cabanov A, Wright RC, Koziol AK, Weiss A, Danahey K, Karrison TG, Edens CC, Bauer Ventura I, Pettit NN, Patel BK, Pisano J, Strek ME, Gajewski TF, Ratain MJ, Reid PD. COVIDOSE: A Phase II Clinical Trial of Low-Dose Tocilizumab in the Treatment of Noncritical COVID-19 Pneumonia. Clin Pharmacol Ther. 2021 Mar;109(3):688-696. doi: 10.1002/cpt.2117. Epub 2020 Dec 10. PMID 33210302

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: Hospitalized, non-critically ill patients with COVID-19 pneumonitis with risk factors for decompensation
  Tocilizumab: Group A: Tocilizumab (beginning dose 200mg) Single dose is provisioned, patient is eligible to receive up to two doses, with re-evaluation of clinical and biochemical responses performed every 24 hours.
  Second dose is provisioned if:
  1. Increasing supplemental oxygen requirement or Tmax higher than baseline in the 24h following initial tocilizumab administration AND
  2. CRP decrease is < 25% at 24 hours following tocilizumab administration and CRP > 40mg/L
- Group B: Hospitalized, non-critically ill patients with COVID-19 pneumonitis without risk factors for decompensation
  Tocilizumab: Group B: Low-dose tocilizumab (beginning dose 80mg) Single dose is provisioned, patient is eligible to receive up to two doses, with re-evaluation of clinical and biochemical responses performed every 24 hours.
  Second dose is provisioned if:
  1. Increasing supplemental oxygen requirement or Tmax higher than baseline in the 24h following initial tocilizumab administration AND
  2. CRP decrease is < 25% at 24 hours following tocilizumab administration and CRP > 40mg/L
Period: Overall Study
Arm/Group | Group A | Group B
Started | 12 | 20
Completed | 12 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 12 | 20 | 32
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 70 [51 to 73] | 66 [41 to 73] | 69 [41 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 11 | 16
  Male | 7 | 9 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 16 | 25
  White | 1 | 0 | 1
  More than one race | 0 | 3 | 3
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 12 | 20 | 32
C-Reactive protein [Mean (Standard Deviation); unit: mg/L] | 175 (83.1) | 138 (76.0) | 152 (79.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Response in Maximum Temperature (Tmax)
Description: Number of Participants with Clinical Response in Maximum Temperature (Tmax)
Time Frame: Assessed for the 24 hour period after tocilizumab administration
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 12 | 20
Participants | 8 | 16

2. Primary Outcome: Number of Participants With Biochemical Response as Determined by CRP Response
Description: Number of Participants with Biochemical Response as determined by CRP Response. Defined as at least 25% decrease in CRP from baseline at least 16 hours after administration of drug.
Time Frame: Assessed every 24 hours during patient's hospitalization, up to 4 weeks after tocilizumab administration
Population: One patient in Group A and 2 patients in Group B were deceased before measure of CRP.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 11 | 18
Participants | 10 | 15

3. Secondary Outcome: Overall Survival
Description: 28-Day Overall Survival is defined as the status of the patient at the end of 28 days, beginning from the time of the first dose of tocilizumab.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 12 | 20
Participants | 10 | 17

4. Secondary Outcome: Survival to Hospital Discharge
Description: This will be defined as the percentage of patients who are discharged in stable condition compared to the percentage of patients who die in the hospital. Patients who are discharged to hospice will be excluded from this calculation.
Time Frame: Hospitalization, up to 4 weeks after tocilizumab administration
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 12 | 20
Participants | 1 | 2

5. Secondary Outcome: Progression of COVID-19 Pneumonitis
Description: This will be a binary outcome defined by worsening COVID-19 pneumonitis resulting in transition from clinical Group A or Group B COVID-19 pneumonitis to critical COVID-19 pneumonitis during the course of the patient's COVID-19 infection. This diagnosis will be determined by treating physicians on the basis of worsening pulmonary infiltrates on chest imaging as well as clinical deterioration marked by persistent fever, rising supplemental oxygen requirement, declining PaO2/FiO2 ratio, and the need for intensive care such as mechanical ventilation or vasopressor/inotrope medication(s).
Time Frame: Hospitalization, up to 4 weeks after tocilizumab administration
Population: No data were collected on this outcome. Given the volumes of patients being cared for and demand for radiology services, it proved impractical during the conduct of the trial to re-examine radiographs of every enrolled patient in the absence of a clinical reason.
Arm/Group | Group A | Group B
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Rate of Non-elective Mechanical Ventilation
Description: This will be a binary outcome defined as worsening COVID-19 disease resulting in the use of non-invasive (BiPap, heated high-flow nasal cannula) or invasive positive pressure ventilation during the course of the patient's COVID-19 infection. For patients admitted to the hospital using non-invasive mechanical ventilation, the utilization of mechanical ventilation will count toward this metric, as well. Calculated as the ratio of the number of patients who require non-invasive or invasive positive pressure ventilation during hospitalization and total number of patients who receive tocilizumab.
Time Frame: Hospitalization, up to 4 weeks after tocilizumab administration
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 12 | 20
Participants | 2 | 4

7. Secondary Outcome: Duration of Mechanical Ventilation
Description: This will be a continuous outcome defined by the amount of time between initiation and cessation of mechanical ventilation (invasive and non-invasive).
Time Frame: Hospitalization, up to 4 weeks after tocilizumab administration
Measure: Median (Full Range); unit: days
Arm/Group | Group A | Group B
Number analyzed (Participants) | 12 | 20
days | 2.5 [0 to 8] | 3.5 [1 to 9]

8. Secondary Outcome: Time to Mechanical Ventilation
Description: This will be a continuous outcome defined by the amount of time between tocilizumab dose administration and the initiation of mechanical ventilation. This will be treated as a time-to-event with possible censoring.
Time Frame: Assessed over hospitalization, up to 4 weeks after tocilizumab administration
Measure: Median (Full Range); unit: days
Arm/Group | Group A | Group B
Number analyzed (Participants) | 12 | 20
days | 2 [0 to 12] | 3.5 [2 to 8]

9. Secondary Outcome: Rate of Vasopressor/Inotrope Utilization
Description: This will be a binary outcome defined as utilization of any vasopressor or inotropic medication during the course of the patient's COVID-19 infection. Calculated as the ratio of the number of patients who require vasopressor or inotrope medication during hospitalization and total number of patients who receive tocilizumab.
Time Frame: Hospitalization, up to 4 weeks after tocilizumab administration
Population: In reviewing inotropic medication utilization, there was a disconnect between orders being placed and medication administration, precluding high-throughput data extraction from electronic health record.
Arm/Group | Group A | Group B
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Duration of Vasopressor/Inotrope Utilization
Description: This will be a continuous outcome defined by the amount of time between initiation of first and cessation of last vasopressor or inotrope medication(s).
Time Frame: Hospitalization, up to 4 weeks after tocilizumab administration
Population: as for outcome 9
Arm/Group | Group A | Group B
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Time to Vasopressor or Inotropic Utilization
Description: This will be a continuous outcome defined by the amount of time between first tocilizumab dose administration and the initiation of vasopressor or inotropic medication(s). This will be treated as a time-to-event with possible censoring.
Time Frame: Assessed over hospitalization, up to 4 weeks after tocilizumab administration
Population: as for outcome 9
Arm/Group | Group A | Group B
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Number of ICU Days
Description: Number of ICU days is defined as the time period when a patient is admitted to the ICU (defined as the timestamp on the first vital signs collected in an ICU) until they are transferred from the ICU to a non-ICU setting such as a general acute care bed (defined as the timestamp on the first vital signs collected outside an ICU, excepting any "off the floor" vital signs charted from operating rooms or procedure or imaging suites). Death in the ICU will be a competing risk.
Time Frame: Hospitalization, up to 4 weeks after tocilizumab administration
Population: Median number of ICU days could not be calculated from our records due to lag in timing of ICU admission order placement, ICU arrival, ICU transfer order, and general ward admission order placement. Therefore, no data was collected for this outcome.
Arm/Group | Group A | Group B
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Duration of Increased Supplemental Oxygen Requirement From Baseline
Description: Duration of increased supplemental oxygen requirement from baseline is defined as the time period (number of days) during which the participant requires supplemental oxygen in excess of his/her baseline supplemental oxygen requirement. The supplemental oxygen requirement is defined as the highest liters-per-minute flow of supplemental oxygen required by the patient each day over the course of the hospitalization.
Time Frame: Assessed over hospitalization, up to 4 weeks after tocilizumab administration
Population: 0 patients analyzed due to heterogeneity in the recording of supplemental oxygen requirement in the electronic health record, complicating data extraction and analysis. There were no patient data collected for this outcome.
Arm/Group | Group A | Group B
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Group A | Group B
All-Cause Mortality (participants affected / at risk) | 2/12 | 3/20
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/20
Other Adverse Events (participants affected / at risk) | 9/12 | 17/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=12) | Group B (N=20)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
QTC prolangulation (Cardiac disorders) | 0 (0) | 1 (1)
Type II NSTEMO (Cardiac disorders) | 1 (1) | 0 (0)
Atrial Flutter (Cardiac disorders) | 0 (0) | 1 (1)
Chest pain (Cardiac disorders) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Blurred vision (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Emisis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Hematoschezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Thick secretions (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1)
Fever (General disorders) | 1 (1) | 1 (1)
Poor appetite (General disorders) | 1 (1) | 1 (1)
H. Pylori infection (Infections and infestations) | 0 (0) | 1 (1)
Acinetobacter PNA (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2)
ALT elevation (Investigations) | 0 (0) | 1 (1)
AST elevation (Investigations) | 0 (0) | 1 (1)
Creatinine elevation (Investigations) | 0 (0) | 1 (1)
BUN elevation (Infections and infestations) | 1 (1) | 0 (0)
Bilirubin elevation (Infections and infestations) | 0 (0) | 1 (1)
Hypokalemia (Endocrine disorders) | 0 (0) | 2 (2)
Starvation ketosis (Endocrine disorders) | 1 (1) | 0 (0)
Hyperglycemia (Endocrine disorders) | 0 (0) | 3 (3)
Hyperkalemia (Endocrine disorders) | 1 (1) | 1 (1)
Hypernatremia (Endocrine disorders) | 0 (0) | 1 (1)
Hypocalcemia (Endocrine disorders) | 0 (0) | 1 (1)
Hypoglycemia (Endocrine disorders) | 0 (0) | 2 (2)
Hypophosphatemia (Endocrine disorders) | 1 (1) | 1 (1)
Transaminitis (Endocrine disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Right arm contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone mineral disease (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Multifocal subacute stroke (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Worsening altered mental status (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 3 (3)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
healthcare-associated pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aspiration event pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Right soleal deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-20): https://cdn.clinicaltrials.gov/large-docs/95/NCT04331795/Prot_SAP_001.pdf